CLINICAL TRIAL: NCT03495583
Title: Effects of Early Introduction of Allergenic Foods Followed by Ad-libitum Consumption, on Food Allergic Sensitisation, Allergy and Measures of Child Health at 8 Years of Age in Exclusively Breastfed Infants
Brief Title: The EAT-On Study: Sensitisation, Allergy and Child Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: King's College London (Other)
Collaborators: Action Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GN2551
Record Dates: First submitted 2018-04-04; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Food Allergy in Children; Obesity, Childhood; Food Allergen Sensitisation
Keywords: Food allergy; Child Health; Oral tolerance induction; Food allergic sensitisation; Obesity
MeSH Terms: conditions — Pediatric Obesity; Food Hypersensitivity; Obesity

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial in which breastfed infants were randomised (equal groups) either to introduce 6 allergenic foods (cow's milk, egg, wheat, peanut, sesame, fish) from 3 months of age or to continue exclusive breastfeeding until about 6 months of age.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early introduction (Experimental): Six commonly allergenic foods introduced (in a randomly assigned order) into the diets of exclusively breastfed infants from about 3 months of age.
  Interventions: Other: Early introduction
- Standard introduction (No Intervention): Infants followed UK DoH standard advice for weaning

INTERVENTIONS:
Other: Early introduction — Consumption of 2g/week of cow's milk, hen's egg, wheat, peanut, sesame and fish protein from 3 months of age (alongside breastfeeding)
  Arms: Early introduction

SUMMARY:
The EAT Study showed a reduction in both sensitisation (to all foods) and clinical food allergy (to peanut and egg) among children who consumed allergenic food early compared with those who followed standard government feeding advice to exclusively consume breast milk for the first 6 months of life. The EAT-On Study aims to establish whether the effects seen at 3 years in the EAT study represent a delay in FA onset or sustained tolerance. EAT-On will also investigate the natural history (emergence and resolution) of FA in childhood; thus shaping dietary and management plans for allergic patients. Findings will inform future research and weaning recommendations for preventing FA.

DETAILED DESCRIPTION:
Sensitisation/Allergy:

Food allergy (FA) is common, increasing in prevalence and represents a public health concern in many countries. FA increasingly affects geographic regions where rates of FA were previously low.(1-5) Data from the Enquiring About Tolerance (EAT) study, which enrolled 1303 exclusively breastfed three month old babies from the general population, showed that 8% of children had proven immediate-onset FA at three years of age. This equates to almost 1 in 10 children. (1) The early-introduction of specific food allergen(s) to infant diets is a successful strategy for the prevention of FA. Introduction of peanut to the infant diet before 11 months of age, protected against the development of peanut allergy in a high-risk, atopic population.(6) This effect persisted despite cessation of peanut consumption for 12 months.(7) In the EAT Study, children from the general population were randomised either to consume six commonly allergenic foods (cow's milk, egg, peanut, wheat, fish and sesame) from four months of age (early introduction group (EIG)), or to follow Department of Health (DoH) advice to exclusively breastfeed until about 6 months of age (standard introduction group (SIG)). The per-protocol analysis revealed a reduction in any FA of 7.3% versus 2.4% (p=0.01), for peanut allergy of 2.5% versus 0% (p=0.003) and for egg allergy 5.5% versus 1.4% (p=0.009) in the SIG and EIG respectively. (8) In the EAT study, between 1 and 3 years an intention-to-treat analysis (ITT) of sensitisation to individual foods showed a significant cumulative treatment effect of 35% (p=0.0095) in the EIG (unpublished data). Furthermore, in the per-protocol analyses (PP), we showed a statistically significant reduction of 41.6% (p=0.01) in skin prick test (SPT) sensitivity to any food at 1 year, and again at 3 years with a 67.3% relative reduction (RR) (p=0.002) in the EIG. These findings were particularly significant for individual food; at 3 years there was a relative reduction in skin-prick sensitivity to all individual foods and particularly for peanut (RR 67.1% p=0.007).

FA is a dynamic condition with egg and milk allergy typically developing in infancy and being outgrown and peanut and sesame allergy usually developing between the ages of 3-6 and persisting into adulthood. Whilst early introduction of commonly allergenic foods is effective in preventing food allergy in early childhood and within the confines of a randomised controlled trial (RCT), the longevity of this novel approach has not been tested and little is known about whether these effects are sustained after 'real world' ad libitum consumption. The EAT-On Study aims to investigate this by following-up children who were previously enrolled in the EAT Study when they are 8 years of age and investigating the natural history of food allergy, and how the intervention that was applied when children were 4-6 months of age influences food allergic sensitisation and clinical food allergy when they are 8 years of age.

Child Health:

Whilst the UK Department of Health recommends exclusive breastfeeding (EBF) until around six months of age, surveys suggest this is achieved by only 1% of mothers(9). Given the lack of EBF till 6 months of age, the majority of infants will require additional nutrition provided from formula and/or solid weaning foods. Indeed, 75% of infants have been introduced to solid food by 5 months of age (9). The nutritional consequences of different weaning regimens may have important consequences on obesity outcomes, but rigorous trials in this area are difficult to undertake, not least because of the necessary ethical concerns that pertain to the comparison of breast-feeding with alternate or complementary feeding strategies. The EAT cohort presents a unique opportunity to study this question further as the diet consumed by children who participated in the EIG of the EAT study is much higher in protein than breastmilk alone. Good quality studies have found that consumption of high protein formula milk in early infancy increases the risk of overweight in later childhood compared with breastfeeding, but the effect of high protein solid food consumption alongside breastfeeding in early infancy has not been studied. The majority of infants have solid food introduced before 6 months of age, and updated guidance advocates the introduction of a high protein food (peanut) from 'around 6 months of age' (UK(10) and Australia(11)), or at 4 months of age (USA(12)) to prevent a new onset of peanut allergy. It is therefore timely to explore how early diet, particularly with respect to high protein weaning diet, influences childhood obesity. This will lead to the development of clearer guidance in respect to early weaning diet which extends to other high protein foods, while taking in to account the risk of childhood obesity.

The nature of the EAT cohort means that between 4 and 6 months of age children were randomised either to a lower protein diet (SIG) or to a higher protein diet (EIG): breastmilk contains approximately 6% energy from protein whilst the EIG were asked to consume a diet containing at least 15% energy from protein, more than double that of the SIG. This cohort therefore offers a unique opportunity to explore the effect of differing energy consumption from dietary protein on overweight/obesity and markers of cardiovascular health in later childhood.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the EAT study
* Age 8 years +/- 12 months

Exclusion Criteria:

* None

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1235 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Allergic sensitisation | 3 years
  Between group differences in total number of cumulative sensitisations to the six study food allergens at age 8
Food allergy | 3 years
  Between group differences in cumulative food allergy (challenge confirmed) t the six study foods at age 8
Child Health | 3 years
  Between group differences in proportion of children who classified as overweight or obese as determined by their BMI and/or BMI z score

SECONDARY OUTCOMES:
Other allergic sensitisations | 3 years
  Between group differences in proportion of children with SPT sensitisation to additional food allergens (hazelnut, brazil nut, cashew, almond and walnut) and aero-allergens (timothy grass, birch pollen, house dust mite, cat and dog dander).
Mechanisms of allergy | 3 years
  Between group differences in specific IgE, IgG and IgG4 to peanut, egg, sesame and aeroallergens
Coeliac disease | 3 years
  Between group differences in prevalence of coeliac disease using coeliac antibody test (tTG IgA) screening test
Atopic dermatitis | 3 years
  Between group differences in prevalence of atopic dematitis
Allergic rhinoconjunctivitis | 3 years
  Between group differences in prevalence of seasonal and perennial rhinoconjunctivitis
Asthma | 3 years
  Between group differences in prevalence of asthma
Oral allergy syndrome | 3 years
  Between group differences in prevalence of oral allergy syndrome
Parent reported food allergy | 3 years
  Between group differences in food reaction history (parent-reported immediate onset food allergy)
Sibling allergies | 3 years
  Prevalence of sibling allergies (food allergies, eczema, asthma and rhinitis)
AGE Level in association with food allergies | 3 years
  Between group differences in AGE levels in association with food allergies
Skin fold thickness | 3 years
  Between group differences in skin fold thickness (triceps and subscapular)
Circumference measurements | 3 years
  Between group differences in midarm, waist and head circumference
Anthropometric ratios | 3 years
  Between group differences in; adjusted weight for height; waist; height ratio; height adjusted weight circumference
Fat free mass | 3 years
  Between group differences in fat free mass
Conicity index | 3 years
  Between group differences in conicity index (calculated from waist circumference and height and weight measurements)
Cardiovascular health | 3 years
  Between group differences in the proportion of children with cardiovascular measurements outside the expected range
Vascular stiffness | 3 years
  Between group differences in vascular stiffness
AGE | 3 years
  Between group differences in advanced glycation end products (AGE)
Inflammation | 3 years
  Between group differences in inflammation (measured using IL=6; sensitive CRP; TNF alpha; MCP-1; RANTES chemokine
Metabolic and endocrine | 3 years
  Between group differences in insulin, IGF-1 and leptin
White cell count | 3 years
  Between group differences in total white blood cell count
Macronutrient dietary intake | 3 years
  Between group differences in macronutrient intake
Dietary habits | 3 years
  Between group differences in fussy eating
Physical activity | 3 years
  Influence of physical activity on anthropometry and body composition measurements
Genetic influences | 3 years
  Influence of parental size on: height; weight; waist circumference on participant's size

CONTACTS AND LOCATIONS:
Locations (1):
- Paediatric Allergy, London, United Kingdom